CLINICAL TRIAL: NCT00455663
Title: Medication Adherence and Outcomes in Schizophrenia
Brief Title: Cognitive Adaptive Training for Improving Medication Adherence, Symptoms, and Function in People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dawn Velligan, Professor, Psychiatry, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH062850 (NIH); R01MH062850 (NIH); DAHBR 96-BHA (Other: UTHSCSA)
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Results first posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Schizophrenia
Keywords: Schizoaffective Disorder; Medication Adherence
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Medication Adherence | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive Adaptation Training (Experimental): In home treatment using environmental supports such as signs, labels, alarms, checklists and the organization of belongings to bypass cognitive impairment, cue and sequence adaptive behavior and improve a wide range of functional outcomes.
  Interventions: Behavioral: Cognitive Adaptation Training
- Pharm-Cognitive Adaptation Training (Experimental): Uses Supports from Cognitive Adaptation Training designed only to promote adherence to medication and treatment follow up.
  Interventions: Behavioral: Pharm-Cognitive Adaptation Training
- Treatment As Usual (Active Comparator): Medication follow up and limited case management provided by local mental health authority
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Cognitive Adaptation Training — Environmental supports for all independent living skills
  Arms: Cognitive Adaptation Training
Behavioral: Pharm-Cognitive Adaptation Training — Environmental supports for medication and appointment adherence
  Arms: Pharm-Cognitive Adaptation Training
Other: Treatment as usual — Medication follow-up and limited case management provided by local community mental health authority
  Arms: Treatment As Usual

SUMMARY:
This study will compare the effectiveness of three treatments in improving medication adherence, symptoms, and function in people with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a chronic and severely disabling mental disorder. People with schizophrenia may experience hallucinations, delusions, disordered thinking, movement disorders, social withdrawal, and cognitive deficits. Antipsychotic medications have been effective in alleviating many of the symptoms of schizophrenia and improving the lives of people with the disease. It is well established, however, that poor adherence to antipsychotic medications can lead to relapse and rehospitalization. Cognitive deficits often contribute to treatment nonadherence by compromising patients' capacity to establish routines for taking medication. Cognitive adaptation training (CAT) is a treatment approach designed to alter the physical environment of individuals with schizophrenia to compensate for cognitive deficits and improve adaptive function. For example, various environmental supports, such as signs, checklists, and electronic devices, are used to remind patients to take their medication. Studies have shown that CAT's support system led to better treatment outcomes than those produced by standard care in people with schizophrenia. This study will compare the effectiveness of two CAT treatments versus standard treatment in improving medication adherence, symptoms, and function in people with schizophrenia.

After providing a blood sample, participants in this single-blind study will be randomly assigned to Full-CAT, Pharm-CAT, or treatment as usual for 9 months. Participants receiving treatment as usual will not receive CAT support. Full-CAT will entail a comprehensive use of environmental supports to improve multiple areas of adaptive functioning. Pharm-CAT will provide support for medication adherence only. Participants assigned to one of the two CAT groups will receive weekly treatments in their homes. All participants will report to the study site once every 3 months to assess medication adherence, symptomatology, and adaptive functioning. Participants will be interviewed by the study physician for 2 to 3 hours at each visit. A member of the study staff will also visit each participant's home at a random, unannounced time once every 3 months to obtain a blood sample. Follow-up visits will occur 3 and 6 months following the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* If entering the study as an inpatient, hospitalization was recent
* Currently receiving treatment with an atypical antipsychotic and continuation on the medication has been recommended
* Assumes primary responsibility for taking medication
* Currently living in a stable environment

Exclusion Criteria:

* History of significant head trauma, seizure disorder, or mental retardation
* History of alcohol or drug abuse or dependence within 1 month prior to study entry
* History of violence within 6 months prior to study entry

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2000-11; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn I. Velligan, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were outpatients recruited in 2 streams. Ninety-nine were recruited at the time of discharge from an inpatient psychiatric facility and followed for 3 months after discharge prior to baseline assessments and randomization
Pre-assignment Details: Of the 99 recruited at hospital Discharge:11 rehospitalized,9 not located,8 withdrew consent,4 incarcerated,3 unable to complete assessments,2 aggressive behavior,2 medication,1 deceased Of 57 outpatient recruits;4 withdrew consent,1 unable to complete assessments,1 medication, 1 unsafe,1 aggression, 1 substance abuse, 1 deceased, 1 moved
Period: Overall Study
Arm/Group | Cognitive Adaptation Training | Pharm-Cognitive Adaptation Training | Treatment As Usual
Started | 37 | 36 | 32
Completed | 34 | 32 | 29
Not Completed | 3 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Adaptation Training | Pharm-Cognitive Adaptation Training | Treatment As Usual | Total
Number analyzed (Participants) | 34 | 32 | 29 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (9.4) | 40 (11.1) | 39 (22.1) | 39.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 11 | 41
  Male | 22 | 14 | 18 | 54

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence-pill Count
Description: % medication taken as determined by unannounced pill counts conducted in the home on 2 occasions in each 3 month period. 1 Final score for endpoint created by averaging scores for 9 months of treatment and 6 months of follow up.
Time Frame: 1 final score combined for endpoint for 9 months of treatment and 6 months follow up
Measure: Least Squares Mean (Standard Error); unit: percentage of medication taken
Groups:
- Pharm-Cognitive Adaptation Training: Environmental supports to assist in medication and appointment adherence
- Treatment as Usual: medication management and case management in the community mental health center
Arm/Group | Pharm-Cognitive Adaptation Training | Cognitive Adaptation Training | Treatment as Usual
Number analyzed (Participants) | 32 | 34 | 29
percentage of medication taken | 80.8 (4.5) | 81.43 (3.7) | 57.3 (3.7)

2. Primary Outcome: Positive Symptoms
Description: Positive symptoms subscale of the Brief Psychiatric Rating Scale includes delusions, hallucinations, conceptual disorganization and suspiciousness-Mean score averaging these items, variability 1-7. Higher scores reflect higher level of symptoms. 1 Final score for endpoint created by averaging scores for 9 months of treatment and 6 months of follow up.
Time Frame: 1 final endpoint least sq mean combining 9 months of treatment 6 months of follow up
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Treatment as Usual: medication management and case management at a community mental health center
Arm/Group | Cognitive Adaptation Training | Pharm-Cognitive Adaptation Training | Treatment as Usual
Number analyzed (Participants) | 34 | 32 | 29
units on a scale | 2.3 (.15) | 2.5 (.17) | 2.3 (.15)

3. Primary Outcome: Social and Occupational Functioning Scale Score
Description: Scores range from 0 to 100 with higher scores reflecting better functioning. 1 Final score for endpoint created by averaging scores for 9 months of treatment and 6 months of follow up.
Time Frame: 1 endpoint ls means combining 9 months of treatment and 6 months follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Adaptation Training | Pharm-Cognitive Adaptation Training | Treatment as Usual
Number analyzed (Participants) | 34 | 32 | 29
units on a scale | 50.8 (1.1) | 45.2 (1.3) | 42.6 (1.2)

4. Primary Outcome: Number of Patients Surviving Without Relapse/Exacerbation
Description: A relapse was scored (only for patients meeting criteria for remission) if scores on any of the 4 items assessing positive symptoms on the Brief Psychiatric Rating Scale increased a minimum of 2 points to a score of 5 or higher, if the patient was suicidal, if the patient was hospitalized, or if the patient was unable to care for themselves without continual supervision
Time Frame: 9 months of treatment 6 months follow up
Population: Number of participants meeting bprs criteria for at least partial remission.scores on 3 of the 4 BPRS psychosis items had to be 4 or lower indicating moderate symptoms only.
Measure: Number; unit: participants
Arm/Group | Cognitive Adaptation Training | Pharm-Cognitive Adaptation Training | Treatment as Usual
Number analyzed (Participants) | 25 | 23 | 21
participants | 15 | 14 | 4

ADVERSE EVENTS:
Time Frame: study duration 15 mos.
Description: Patient reported events
Arm/Group | Cognitive Adaptation Training | Pharm-Cognitive Adaptation Training | Treatment As Usual
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32 | 0/29
Other Adverse Events (participants affected / at risk) | 0/34 | 0/32 | 0/29

LIMITATIONS AND CAVEATS:
Subjects were ill for a long-period of time

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No